CLINICAL TRIAL: NCT05389592
Title: Treatment of COVID-19 Post-acute Cognitive Impairment Sequelae (PASC) With Portable Brain Stimulation: a Double-blind, Randomized-controlled Trial
Brief Title: Treatment of COVID-19 Post-acute Cognitive Impairment Sequelae With tDCS
Acronym: PASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Andre R Brunoni, Associate Professor of the Medical School of the University of Sao Paulo (FMUSP), Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 52917821.1.0000.0068
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Impairment; Post-Acute Sequelae of SARS-CoV-2 Infection; COVID-19
MeSH Terms: conditions — Cognitive Dysfunction; Post-Acute COVID-19 Syndrome; COVID-19 | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Double-active (Experimental): Active transcranial electrical stimulation and cognitive training.
  Interventions: Procedure: Active tDCS and cognitive training
- Cognitive training-only (Sham Comparator): Sham transcranial electrical stimulation and cognitive training.
  Interventions: Procedure: Sham tDCS and cognitive training

INTERVENTIONS:
Procedure: Active tDCS and cognitive training — Electrical stimulation is delivered by the Soterix device, consisting of a one-size-fits-all, transcranial direct current stimulation headset with square electrodes. The anode is positioned over the left prefrontal cortex, and the cathode over the right prefrontal cortex. Current strenght is set at 2mA for 20 minutes, daily for 5 continuous days (with a 2-day pause) for 4 weeks. Cognitive training consists of a series of tasks performed in the BrainHQ app, which aim to stimulate the impaired cognitive domains in people with PASC. The cognitive training sessions are performed concomitantly to the tDCS sessions.
  Arms: Double-active
Procedure: Sham tDCS and cognitive training — Sham electrical stimulation is delivered by the Soterix device, consisting of a one-size-fits-all, transcranial direct current stimulation headset with square electrodes. The anode is positioned over the left prefrontal cortex, and the cathode over the right prefrontal cortex. The sham protocol consists of a fade-in and fade-out phases of 1mA for 45 seconds, followed by a silent period in between for the remaining session time. Cognitive training consists of a series of tasks performed in the BrainHQ app, which aim to stimulate the impaired cognitive domains in people with PASC. The cognitive training sessions are performed concomitantly to the tDCS sessions.
  Arms: Cognitive training-only

SUMMARY:
After almost 2 years of pandemic, the consequences of the post-COVID syndrome, or PASC (Post Acute-Sequelae of Sars-CoV-2), have become a major challenge in the management of affected patients, generating costs for health services. and insecurity regarding treatments for the sequelae, given the complex and still poorly understood pathophysiology of COVID-19.

This troubling scenario raises important questions about the impact of COVID-19 on central nervous system sequelae, including the risk of cognitive decline in old age and progression to dementia. Therefore, studies that propose the possibility of treatment for this new clinical condition and that are free from systemic side effects, such as transcranial direct current stimulation (tDCS) and cognitive treatment, are extremely important in the face of this scenario. In addition, the evaluation of the neural mechanisms underlying the cognitive alterations of the PASC syndrome and after the treatment using multimodal magnetic resonance imaging (MRI) becomes relevant in view of the lack of studies related to the topic.

Therefore, the objective of this double-blind randomized clinical trial is to assess whether tDCS associated with cognitive training can improve symptoms in patients with persistent cognitive deficits that started between 1 and 6 months after the resolution of acute COVID-19 infection (PASC) compared to the sham (placebo) group, in addition to exploring the structural, microstructural, functional and modeled electric field changes associated with cognitive alterations due to PASC syndrome and tDCS combined with cognitive treatment. 60 patients aged between 18 and 70 years and with a positive diagnosis of mild to moderate COVID-19 in the last 6 months in relation to the time of entry into the study will be recruited. All of them will be pre-screened online and in person to confirm the cognitive dysfunction associated with PASC.

DETAILED DESCRIPTION:
As of August 1, 2021, novel coronavirus disease 2019 (COVID-19), an infection caused by Severe Acute Respiratory Syndrome (SARS-CoV-2), had infected over 200 million people and accounted for more than 4 million deaths worldwide. After remission of the acute phase of the disease, many patients report persistent symptoms that go far beyond the consequences of the pulmonary involvement itself and can impose chronic sequelae of COVID-19. According to the World Health Organization, post-COVID-19 syndrome occurs in individuals with a history of probable or confirmed SARS CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms and lasting at least 2 months and cannot be explained by an alternative diagnosis. The most common complaints are extreme fatigue, inability to perform activities of daily living that involve physical or cognitive exertion, emotional dysregulation, mental fog, and other symptoms of cognitive impairment. Symptoms may be new after initial recovery from an acute episode of COVID-19 or persist from the initial illness. Symptoms can also fluctuate or recur over time.

Given the increasing number of COVID-19 cases, there is an urgent need to develop treatment alternatives for PASC-related cognitive and memory deficits. In this context, transcranial direct current stimulation (tDCS or tDCS) is a non-invasive brain stimulation intervention that may be promising in these cases. It represents an interesting opportunity for targeting the neural circuits underlying neurological, cognitive, and psychiatric disorders. For example, once a target neural circuit has been identified as a related region of interest for a neuropsychiatric disorder, neuromodulation methods could be used to selectively modify activities in the target region. In tDCS, a direct, low-intensity electrical current (e.g., typically 1-4 mA) is passed through at least two electrodes (i.e., anode and cathode), which are applied non-invasively to the scalp. TDCS modulates neuronal activity at the network level by producing current flow around neurons and resulting in an incremental change in neuronal membrane potentials. In turn, such potential changes lead to a series of changes in neuronal function, such as a change in firing rates.

Thus, tDCS can induce long-term changes in brain activity. Learning ability requires functional changes that can be induced by tDCS, which makes this technique a promising tool to improve cognitive performance. In fact, tDCS has already been successfully used in non-COVID-19 samples to improve cognitive performance in several domains, such as working memory, episodic memory, executive function, and language. It is also worth noting that tDCS presents definite or probable evidence of efficacy for several neuropsychiatric disorders that are often accompanied by cognitive deficits such as addiction, attention deficit/hyperactivity disorder, Parkinson's disease (motor and cognitive impairment), epilepsy, schizophrenia, Alzheimer's disease, and depression.

TDCS has attractive advantages for clinical use, such as affordability, lower cost than magnetic stimulation, ease of use and operation, especially for customized devices, and portability. In fact, the development of portable devices with remote control allows for greater ease of use and feasibility in uncontrolled pandemic scenarios. Furthermore, recent evidence suggests that the effects of tDCS may be enhanced by a concomitantly administered intervention. Neurophysiological studies have shown that tDCS parameters used in clinical practice have an unlikely impact on neural spiking, as such modulation is only achieved at doses ≥ 4.5mA. Rather, the effects of tDCS on behavior are best explained by modulating ongoing activity. According to the "selective activity" hypothesis, tDCS preferentially modulates a neuronal network that is already activated, rather than separate inactive neuronal networks. For example, in vitro direct current stimulation (DCS) preferentially increased plasticity in a synaptic pathway previously stimulated at 0.1 Hz, whereas DCS alone, without preactivation, did not influence synaptic efficacy. Another study showed that anodic DCS increased long-term potentiation (LTP) induced by high-frequency stimulation, but did not induce LTP per se. In other words, preclinical studies have shown that tDCS is too nonspecific to alter synaptic efficacy alone, but can enhance Hebbian (associative) plasticity activated by task performance.

The pupillary light reflex (PLR) is a reflex that controls the diameter of the pupil in response to variations in light intensities that reach the retina and is modulated by the autonomic nervous system (ANS) that innervate the circular and radial muscles of the iris, while contracting or relaxing, decrease or increase the size of the pupil, respectively. Studies have shown that a specific selection of intensity and light stimulus, wavelength and duration directly influence the contributions of retinal photoreceptors, making it possible to also assess retinal changes beyond the ANS. Patients with Alzheimer's Disease (AD) are known to have alterations in cholinergic neurotransmission, in a decrease in pupil diameter response to abrupt changes in room lighting or a single flash of light. Therefore, the RPL is a good tool for evaluating patients with AD.

Another potentially relevant change may occur in the regulation of the ANS in the heart rate, which can be measured by checking the heart rate variability (HRV). This type of measurement involves the collection of HR for approximately 5 minutes, allowing measurements in the frequency domain, being separated into two bands: the high frequency, associated with vagal activity, and the low frequency, associated with sympathetic activity. There is evidence that HRV is decreased in several cognitive disorders. Thus, it is reasonable to assume that the HRV may also be altered in the PASC. In fact, a point of convergence between AD and the cognitive sequelae of COVID-19 would be precisely autonomic dysfunction - chronic, progressive and of neurodegenerative etiology in the case of AD, and acute, caused by the "inflammatory storm" of COVID-19 and its multisystem consequences. Thus, the investigation of this biomarker can help in the understanding of cognitive PASC.

MRI assessments have become important in the study of brain structure and function, their respective changes and associations with clinical and neuropsychological assessment scores. Neuroimaging studies on COVID-related pathologies and associations with cognitive changes, in addition to the assessment of the impacts of non-invasive brain stimulation, are embryonic. Reviews of acute and chronic effects have been published, although they are more qualitative in terms of the damage caused, without exploring quantitative markers of brain structure, microstructure and function. Therefore, the present project is a pioneer in identifying alterations in quantitative markers of multimodal MRI, their associations with neuropsychological assessment scores and for evaluating the effects of tDCS combined with cognitive treatment in a group of patients with CSBP.

The aim of this double-blind randomized clinical trial is to assess whether tDCS combined with cognitive training can improve symptoms in patients with persistent cognitive deficits that started between 1 and 6 months after resolution of acute COVID-19 infection (PASC or syndrome of long-covid) compared to the sham (placebo) group.

In addition, it is aimed to describe the subjective symptoms related to PASC; to assess whether the RPL is altered in patients with post-COVID cognitive impairment and whether it can be used as a biomarker for treatment response; to assess whether HRV is altered in patients with post-COVID cognitive impairment and whether it can be used as a biomarker for treatment response; to evaluate the neural mechanisms underlying the cognitive alterations of the PASC syndrome; and to assess brain changes after tDCS treatment combined with cognitive treatment using multimodal magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 70 years;
* Positive diagnosis (confirmed by RT-PCR nasal swab) of COVID-19 within the last 6 months in relation to the time of assessment;
* Mild to moderate COVID-19 disease (no hospital stay required);
* A score above 10 in the cognitive symptoms domain of the Post-COVID-19 Symptom Assessment Questionnaire;
* Clinical neuropsychological assessment/neurological examination indicating cognitive impairment after acute COVID illness.

Exclusion Criteria:

* Contraindications to the use of tDCS (such as metal plates on the head);
* Severe acute COVID-19 illness;
* Less than 8 years of schooling;
* Presence of serious neurological conditions such as neurocognitive disorders, stroke, lacunar infarction, cerebral atrophy and others;
* Presence of serious psychiatric disorders, such as untreated mood disorders (including suicidal ideation), personality disorders, or psychotic disorders;
* Unstable clinical conditions;
* Use of medications (such as benzodiazepines and anticonvulsants) that can impair cognition;
* Presence of pathological neuroimaging findings (eg, acute or subacute lacunar or hemorrhagic stroke and others);
* Presence of a pacemaker, orthosis or prosthesis incompatible with the performance of magnetic resonance imaging;
* Claustrophobia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Change in neuropsychological assessment between experimental groups | Week 0 (baseline) and Week 4 (endpoint)
  A battery of neuropsychological tests to assess memory, attention, executive functions and mood.

SECONDARY OUTCOMES:
Change in pupillary reflex | Week 0 (baseline) and Week 4 (endpoint)
  Roland system, composed of a Ganzfeld (Roland Consult), with light-emitting diodes responsible for the stimulus and an infrared camera, capable of recording images in the dark with high spatial and temporal resolution, in continuous recording in recording mode at 30 Hz
Brain changes using multimodal magnetic resonance imaging (MRI) | Week 0 (baseline)
  Functional and structural MRI scans
Change in heart rate variability (HRV) between experimental groups | Week 0 (baseline) and Week 4 (endpoint)
  Heart rate measure with Polar device

CONTACTS AND LOCATIONS:
Overall Officials: André R Brunoni, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Instituto de Psiquiatria, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charvet L, Shaw M, Dobbs B, Frontario A, Sherman K, Bikson M, Datta A, Krupp L, Zeinapour E, Kasschau M. Remotely Supervised Transcranial Direct Current Stimulation Increases the Benefit of At-Home Cognitive Training in Multiple Sclerosis. Neuromodulation. 2018 Jun;21(4):383-389. doi: 10.1111/ner.12583. Epub 2017 Feb 22. PMID 28225155
- [Background] Charvet LE, Yang J, Shaw MT, Sherman K, Haider L, Xu J, Krupp LB. Cognitive function in multiple sclerosis improves with telerehabilitation: Results from a randomized controlled trial. PLoS One. 2017 May 11;12(5):e0177177. doi: 10.1371/journal.pone.0177177. eCollection 2017. PMID 28493924
- [Background] Eilam-Stock T, George A, Charvet LE. Cognitive Telerehabilitation with Transcranial Direct Current Stimulation Improves Cognitive and Emotional Functioning Following a Traumatic Brain Injury: A Case Study. Arch Clin Neuropsychol. 2021 Apr 21;36(3):442-453. doi: 10.1093/arclin/acaa059. PMID 33885138
- [Background] Kim PH, Kim M, Suh CH, Chung SR, Park JE, Kim SC, Choi YJ, Lee JH, Kim HS, Baek JH, Choi CG, Kim SJ. Neuroimaging Findings in Patients with COVID-19: A Systematic Review and Meta-Analysis. Korean J Radiol. 2021 Nov;22(11):1875-1885. doi: 10.3348/kjr.2021.0127. Epub 2021 Jul 1. PMID 34269530
- [Background] Dedoncker J, Brunoni AR, Baeken C, Vanderhasselt MA. A Systematic Review and Meta-Analysis of the Effects of Transcranial Direct Current Stimulation (tDCS) Over the Dorsolateral Prefrontal Cortex in Healthy and Neuropsychiatric Samples: Influence of Stimulation Parameters. Brain Stimul. 2016 Jul-Aug;9(4):501-17. doi: 10.1016/j.brs.2016.04.006. Epub 2016 Apr 12. PMID 27160468
- [Background] Baptista AF, Baltar A, Okano AH, Moreira A, Campos ACP, Fernandes AM, Brunoni AR, Badran BW, Tanaka C, de Andrade DC, da Silva Machado DG, Morya E, Trujillo E, Swami JK, Camprodon JA, Monte-Silva K, Sa KN, Nunes I, Goulardins JB, Bikson M, Sudbrack-Oliveira P, de Carvalho P, Duarte-Moreira RJ, Pagano RL, Shinjo SK, Zana Y. Applications of Non-invasive Neuromodulation for the Management of Disorders Related to COVID-19. Front Neurol. 2020 Nov 25;11:573718. doi: 10.3389/fneur.2020.573718. eCollection 2020. PMID 33324324
- [Derived] Vidal KS, Cavendish BA, Goerigk S, Pita Batista M, Oliveira Lima AR, Pinto BS, Neto Domingos AA, de Sousa JP, Pelosof R, Bertola L, Silva V, Suemoto CK, Razza LB, Bikson M, Pilloni G, Charvet L, Silva PHR, Brunoni AR. Transcranial direct current stimulation plus cognitive training for cognitive symptoms in patients with post-acute sequelae of SARS-CoV-2 infection: A randomized, double-blind, sham-controlled trial. Brain Stimul. 2025 Sep-Oct;18(5):1608-1616. doi: 10.1016/j.brs.2025.08.018. Epub 2025 Aug 21. PMID 40848897